CLINICAL TRIAL: NCT01913795
Title: Environmental Intervention to Reduce Allergens in Urban Schools and Childhood Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Wanda Phipatanakul, Associate Professor of Pediatrics, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 266134
Record Dates: First submitted 2013-05-21; First posted 2013-08-01 (Estimated); Results first posted 2015-10-14 (Estimated); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Air Filters

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Environmental Intervention (Active Comparator): 4 classroom air purifiers and school integrated pest management environmental intervention
  Interventions: Other: integrated pest management; Other: air purifier
- Sham and Control (Placebo Comparator): 4 sham air purifiers and no school integrated pest management environmental intervention
  Interventions: Other: Sham air purifier
- Active Air Purifier and Control (Placebo Comparator): 4 air purifiers and no school integrated pest management environmental intervention
  Interventions: Other: air purifier
- Sham and Integrated Pest Management (Sham Comparator): 4 classroom sham air purifiers and school integrated pest management
  Interventions: Other: integrated pest management

INTERVENTIONS:
Other: integrated pest management — integrated pest management and environmental strategy
  Arms: Environmental Intervention; Sham and Integrated Pest Management
Other: air purifier — air purifiers
  Arms: Active Air Purifier and Control; Environmental Intervention
Other: Sham air purifier — sham air purifiers
  Arms: Sham and Control

SUMMARY:
The investigators aim to pilot the role of school based intervention consisting of enhanced integrated pest management, classroom air purifiers and cleaning improves asthma morbidity.

DETAILED DESCRIPTION:
By piloting this school based intervention, the investigators hope to learn from this study the best way to design and implement more cost and time efficient large-based school-based environmental interventions that may potentially help a community of children with asthma, allergic diseases, and its associated morbidity.

ELIGIBILITY:
Inclusion Criteria:

* grades K-8 with asthma attending sampling/intervention schools

Exclusion Criteria:

* moving schools

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2013-05; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Air Purifier + IPM: classroom air purifiers and school integrated pest management environmental intervention
  integrated pest management: integrated pest management and environmental strategy
  air purifier: air purifiers
- Sham and no IPM: sham air purifiers and no school integrated pest management environmental intervention
- Air Purifier and no IPM: air purifiers and no school integrated pest management environmental intervention
  air purifier: air purifiers
- Sham and IPM: classroom sham air purifiers and school integrated pest management
  integrated pest management: integrated pest management and environmental strategy
Period: Overall Study
Arm/Group | Air Purifier + IPM | Sham and no IPM | Air Purifier and no IPM | Sham and IPM
Started | 4 | 10 | 9 | 6
Completed | 4 | 7 | 9 | 5
Not Completed | 0 | 3 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Air Purifier + IPM | Sham and no IPM | Air Purifier and no IPM | Sham and IPM | Total
Number analyzed (Participants) | 4 | 7 | 9 | 5 | 25
Age, Continuous [Mean (Full Range); unit: years] | 8.6 [7 to 10] | 10.0 [8 to 12] | 9.2 [7 to 11] | 9.4 [8 to 12] | 9.4 [7 to 12]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6 | 3 | 15
  Male | 2 | 3 | 3 | 2 | 10
Forced Vital Capacity (FVC) [Mean (Full Range); unit: Liters] | 1.4 [1.2 to 1.7] | 1.6 [.8 to 2.5] | 1.6 [1.1 to 2.3] | 1.8 [1.2 to 2.4] | 1.6 [.8 to 2.5]

OUTCOME MEASURES:

1. Primary Outcome: Asthma Symptoms
Description: number of days of wheezing/cough
Time Frame: over a two week period at Baseline and Months 3, 6, 9 and 12
Population: The number of participants analyzed here excludes participants for whom follow-up for health outcomes was incomplete.
Measure: Mean (Full Range); unit: Days
Groups:
- Air Purifier + IPM: 4 subjects
  classroom air purifiers and school integrated pest management environmental intervention
  integrated pest management: integrated pest management and environmental strategy
  air purifier: air purifiers
- Sham and no IPM: 7 subjects
  sham air purifiers and no school integrated pest management environmental intervention
- Air Purifier and no IPM: 9 subjects
  air purifiers and no school integrated pest management environmental intervention
  air purifier: air purifiers
- Sham and IPM: 5 subjects
  classroom sham air purifiers and school integrated pest management
  integrated pest management: integrated pest management and environmental strategy
Arm/Group | Air Purifier + IPM | Sham and no IPM | Air Purifier and no IPM | Sham and IPM
Number analyzed (Participants) | 4 | 7 | 9 | 5
Days
  baseline | 1.5 [0 to 3] | 2.9 [0 to 14] | 1 [0 to 3] | 0.4 [0 to 2]
  month 3 | 5.5 [2 to 9] | 7.3 [0 to 14] | 1.3 [0 to 2] | 2.7 [2 to 4]
  month 6 | 5 [5 to 5] | 3.25 [0 to 5] | 2 [2 to 2] | 0.5 [0 to 1]
  month 9 | 3.5 [3 to 4] | 8.25 [2 to 14] | 2.5 [0 to 5] | 1.5 [0 to 3]
  month 12 | 14 [14 to 14] | 1 [1 to 1] | 1.3 [0 to 2] | 0 [0 to 0]

2. Secondary Outcome: Lung Function
Description: peak expiratory flow (PEF)
Time Frame: measured at baseline and months 6 and 12
Population: The number of participants analyzed here excludes participants for whom follow-up for health outcomes was incomplete.
Measure: Mean (Standard Error); unit: Liters/second
Arm/Group | Air Purifier + IPM | Sham and no IPM | Air Purifier and no IPM | Sham and IPM
Number analyzed (Participants) | 4 | 7 | 9 | 5
Liters/second
  Baseline | 3.1 (0.3) | 2.9 (0.3) | 2.7 (0.4) | 3.6 (0.3)
  month 6 | 3.1 (0.3) | 3.3 (0.5) | 2.9 (0.3) | 3.7 (0.3)
  month 12 | 3.1 (0.5) | 3.3 (0.5) | 3.3 (0.3) | 4.0 (0.7)

ADVERSE EVENTS:
Arm/Group | Air Purifier + IPM | Sham and no IPM | Air Purifier and no IPM | Sham and IPM
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/7 | 0/9 | 0/5
Other Adverse Events (participants affected / at risk) | 0/4 | 0/7 | 0/9 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No